CLINICAL TRIAL: NCT01444300
Title: Dalfampridine to Improve Imbalance in Multiple Sclerosis: A Pilot Study
Brief Title: Dalfampridine for Imbalance in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Acorda Therapeutics (Industry)
Responsible Party: Principal Investigator, Michelle Cameron, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNEUR0637A
Record Dates: First submitted 2011-09-20; First posted 2011-09-30 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: multiple sclerosis; postural balance; gait; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dalfampridine (Experimental)
  Interventions: Drug: Dalfampridine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalfampridine — 10mg, bid, pill taken by mouth for 12 weeks
  Other Names: Ampyra
  Arms: Dalfampridine
Drug: Placebo — placebo pill, bid for 12 weeks
  Arms: Placebo

SUMMARY:
Dalfampridine is a new medication that was FDA approved in 2010 to improve walking speed in people with Multiple Sclerosis (MS). People with MS walk slowly in part because MS damages the myelin insulation around nerves which slows conduction of messages from the brain to the leg muscles. Dalfampridine works by improving conduction in nerves with damaged myelin. Recent research indicates that imbalance in MS is in large part caused by poor conduction by the nerves that transmit information about the position of the legs to the brain. It is therefore likely that, by improving nerve conduction, dalfampridine will also improve imbalance in people with MS. Dalfampridine will be administered in this study by the same route (oral), dosage (10mg), and frequency (every 12 hours) approved by the FDA to improve walking speed in people with MS. The proposed pilot study will examine the effects of dalfampridine on imbalance in 24 subjects with Multiple Sclerosis (MS) and imbalance. This small pilot study will help to show if dalfampridine improves imbalance in MS and will guide the design and implementation of a larger full scale study to definitively determine if dalfampridine improves balance and prevents falls in people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Age 20- 59 years,
* Able to walk at least 100m without an aide or with unilateral assistance
* Prolonged APR latencies (≥ 1SD > mean for healthy people in this age range) OR,
* Reduced balance-related activity (ABC scores ≤ 85%),
* Abnormal trunk range of motion (horizontal), trunk range of motion (frontal), turning duration, cadence, double support time, stride length or gait cycle time (outside 1SD of the average for healthy people in this age range)

Exclusion Criteria:

* Currently taking dalfampridine (any within the last 2 weeks),
* Cause(s) of imbalance other than MS,
* Impaired renal function (creatinine clearance ≤50mL/min),
* Seizure disorder
* Pregnancy or breast feeding

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: OHSU Multiple Sclerosis Center — http://www.ohsu.edu/ms

RESULTS

PARTICIPANT FLOW:
Recruitment Details: People with MS were recruited from several MS clinics in the Portland, OR metro area from September 2011 to August 2013. 24 subjects signed the consent and were enrolled in the study.
Groups:
- Dalfampridine: Dalfampridine: 10mg, twice daily, pill taken by mouth for 12 weeks
- Placebo: Placebo: placebo pill, twice daily, for 12 weeks
Period: Overall Study
Arm/Group | Dalfampridine | Placebo
Started | 12 | 12
Completed | 8 | 12
Not Completed | 4 | 0
Not completed — Adverse Event | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dalfampridine: Dalfampridine: 10mg, twice daily (bid), pill taken by mouth for 12 weeks
- Placebo: Placebo: placebo pill, twice daily (bid), for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Dalfampridine | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (8.9) | 47.8 (10.9) | 47.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
MS Subtype [Number; unit: participants]
  Relapsing Remitting MS (RRMS) | 12 | 8 | 20
  Secondary Progressive MS (SPMS) | 0 | 2 | 2
  Primary Progressive MS (PPMS) | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Automatic Postural Response (APR )Latency
Description: Automatic Postural Response (APR) latencies will be measured by Computerized Dynamic Posturography (CDP). The restoration of balance after an unexpected movement by Computerized Dynamic Posturography relies on automated postural responses in the upper and lower legs, trunk, shoulders, and neck muscles. APR latency is the reaction- time response to movements of the support surface on which the subject stands. These responses typically occur at onset latencies of ~100 milliseconds. In response to a change, both feet-in-place and stepping strategies can be used to recover balance, with the incidence of stepping responses becoming larger as the change magnitude increases voluntary movements in human subjects.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Placebo: Placebo: placebo pill, twice daily (bid), pill taken by mouth for 12 weeks
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 8 | 12
milliseconds | 5.71 (16.2) | 4.58 (23.0)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; t test comparing change in outcome between active and placebo; Test type: Superiority or Other; p = 0.51, t-test, 2 sided

2. Secondary Outcome: Change in Activities-specific Balance Confidence (ABC) Questionnaire Scores
Description: The ABC is an 11-point scale and subjects are asked to indicate personal level of confidence in doing specific activities without losing balance or becoming unsteady on a scale from 0% to 100%. The ratings are added (possible range =0 -1600) and divide by 16 to get each subject's ABC score. A high ABC score indicates a high degree of confidence and a low ABC score indicates a low degree of confidence.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 8 | 12
Scores on a scale | 1.30 (9.02) | 0.41 (10.7)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; t test comparing change in outcome between active and placebo after 12 weeks; Test type: Superiority or Other; p = 0.7, t-test, 2 sided

3. Secondary Outcome: Change in Timed 25 Foot Walking Speed
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Placebo: Placebo: placebo pill, twice daily (bid), pill taken by mouth for for 12 weeks
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 8 | 12
seconds | 0.26 (0.78) | 0.39 (1.45)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; t test comparing change in outcome between active and placebo; Test type: Superiority or Other; p = 0.8, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Dalfampridine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/12 | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalfampridine (N=12) | Placebo (N=12)
Insomnia (Nervous system disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Balance problems (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Itching/skin reactions (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less